CLINICAL TRIAL: NCT02021162
Title: Open-label, Single-blinded, Observational, Prospective, 24-months, Longitudinal, Controlled Study to Assess the Efficacy of Gilenya® on Development of Thalamus Pathology and Cognitive Impairment in Patients With Relapsing Forms of Multiple Sclerosis.
Brief Title: Effects of Gilenya (Fingolimod) on Thalamus Pathology and Cognitive Impairment in Patients With Relapsing Forms of Multiple Sclerosis
Acronym: GLT
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, Director, Buffalo Neuroimaging Analysis Center, Professor, University at Buffalo
Other Study IDs: Gilenya-thalamus
Record Dates: First submitted 2013-12-19; First posted 2013-12-27 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Multiple Sclerosis; Healthy
Keywords: Multiple sclerosis; Gilenya; Healthy controls; Thalamic atrophy; MRI
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gilenya: MS patients taking Gilenya
- Healthy Controls: Healthy controls age and gender matched to MS patients taking Gilenya

SUMMARY:
This study aims to assess the effect of Gilenya on brain pathology and cognitive impairment over 6, 12, and 24 months in patients with relapsing MS using MRI, clinical data, and neurological assessments. Healthy controls will also be followed over 6, 12, and 24 months using the same measures.

DETAILED DESCRIPTION:
This is an open-label, single-blinded, observational, prospective, 24 months follow-up, controlled study to assess the efficacy of Gilenya on thalamus pathology and cognitive impairment in 30 relapsing MS patients naïve to Gilenya who fulfilled the inclusion and exclusion criteria used for screening and started Gilenya, on a clinical basis. In addition, 20 HCs will be included as a reference population. Because this is an observational study investigating evolution of thalamic atrophy, iron deposition, cognitive dysfunction and response to herpes viruses in patients treated with Gilenya on a clinical basis the patients are not starting Gilenya as an investigational drug. Therefore, the patients who are already started Gilenya by the treatment decision of their physician will be asked to participate in this observational study.

The screening and starting procedures criteria for Gilenya on a clinical basis and for our study are defined by the Gilenya PI. All patients in our clinic have standardized assessments before starting any disease-modifying therapy. Once the patient decided to start Gielnya on a clinical basis and qualified on a screening, as defined by Gilenya PI, our team will be informed and contact the patient regarding participation in the present study before receiving first dose of Gilenya. Once the informed consent is signed, the patient will follow study procedures, as outlined in the protocol and study evaluation schedule. All subjects will be assessed at 0, 6, 12 and 24 months with the same clinical, 3T MRI and laboratory, and humoral response to herpes viruses examinations. The cognitive assessments and evaluation of environmental risk factors will be performed at 0, 12 and 24 months. Safety will be also assessed at 0, 6, 12 and 24 months of the study.

The healthy controls (HC) will serve as reference comparison group to patients for atrophy iron, cognitive and response to herpesvirus outcomes. We considered alternative study designs as listed below. The head-to-head comparison with untreated or comparator-treated patients are difficult to conduct and can not be performed without proper randomization and double-blinding which is costly and unfeasible in mechanistical study like is the one proposed. The inclusion of a HC group provides a valuable baseline, allowing evaluation of the proposed techniques for normal variation between individuals, against which changes in the proposed outcomes could be compared. Use of HCs for comparison with a patient population in prospective longitudinal pilot studies of non-conventional MRI, including measurement of thalamic atrophy and iron deposition, may become an attractive approach in the future for several reasons. First, the ultimate goal of therapy is to normalize patient changes over time, to those observed in HCs over the same time period. HCs also experience brain changes over time and so the notion of arresting disease progression as measured by proposed outcomes requires validation by reference to a comparator without disease progression to account for age-related changes. Second, ethical considerations preclude placebo-controlled studies using an established MS treatment versus placebo-treatment in patients with RRMS.

The MRI analysis will be performed fully blinded, as are all phase I, II, III and IV trials calculated at the Buffalo Neuroimaging Analysis Center (BNAC), Buffalo, NY. BNAC has been involved as an centralized MRI reading center in many MS clinical trials that included over 500 sites around the world in 55 countries The detailed procedures of how the MRI DICOM files are blinded and how the workload is distributed are part of our internal standard operating procedures (SOPs) that have been accepted as appropriate following standard audits by government and industry agencies.

All participants will undergo study eligibility screening and consenting by a Clinical Research Project Coordinator. The participant will be provided with a description of the required testing for study participation, and any risks will be described in order for the person to make an informed decision regarding voluntary study participation. This is also an opportunity for the person to ask questions regarding the study and the testing components. All study participants who choose to enroll in the study will be asked to sign and date the consent form in front of the Study Coordinator who will also sign and date the consent as witness.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with MS according to McDonald criteria
* Age 18-60
* Have a relapsing disease course or a Healthy Control
* Have EDSS scores 0-6.5
* Have a disease duration <20 years
* Patients who have been clinically cleared and have agreed with their neurologist to begin therapy with Gilenya will be asked to enroll in this prospective study. No drug will be administered as part of this study.
* Be willing and able to comply with the study procedures for the duration of the trial
* Have given written informed consent and signed Health Insurance Portability and Accountability Act (HIPAA) Authorization before any study-related activities are carried out
* Normal kidney functioning (creatinine clearance >59) - patients only
* None of the exclusion criteria

Exclusion Criteria:

* Have received treatment within 30 days prior to enrollment with steroids or any other concomitant immunomodulatory therapies (e.g., interferon-beta, glatiramer acetate, intravenous immunoglobulin)
* Less than 6 months from the use immunosuppressant agents (e.g. including but not limited to mitoxantrone, cyclophosphamide, azathioprine, methotrexate, CellCept, natalizumab
* Ever use of cladribine, fludarabine, or total body irradiation) alemtuzumab/Campath
* Have received an investigational drug or experimental procedure within the past 30 days
* Women who are pregnant, lactating or of childbearing age who do not consent to approved contraceptive use during the study
* Abnormal blood tests (pre-dose assessment as per site procedure for patients considered for Gilenya treatment), including ALT or AST greater than two times the upper limit of normal

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 30 relapsing MS patients naïve to Gilenya who fulfill the inclusion and exclusion criteria used for screening and start Gilenya, on a clinical basis will be enrolled in the study. In addition, 20 healthy controls will be included as a reference population. The plan is to recruit the 50 subjects (30 relapsing MS and 20 healthy controls) at a single center.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-11; Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Thalamic atrophy | 6, 12, and 24 months
  To assess the effect of the Gilenya over 6, 12 and 24 months on the evolution of thalamic atrophy in patients with relapsing MS, as measured by change in thalamic volume loss. The changes in thalamic volume over the same time period in HC will be used as a reference.

SECONDARY OUTCOMES:
Thalamic pathology | 6, 12, and 24 months
  To examine the effect of the Gilenya over 6, 12 and 24 months on the evolution of thalamic pathology in patients with relapsing MS, as measured by change in MP-LPV. The changes in MP-LPV of the thalamus over same time period in HC will be used as a reference.
Cognitive impairment | 12 and 24 months
  To determine the effect of the Gilenya over 12 and 24 months on the evolution of cognitive impairment in patients with relapsing MS, as measured by changes in Minimal Assessment of Cognitive Function (MACFIMS) battery. The cognitive changes over the same time period will be examined in HC, and used as a reference.
Thalamic volume and accumulation of iron in response to herpes viruses | 24 months
  To investigate the association between development of thalamus pathology, as defined by changes in thalamic volume loss and accumulation of MP-LPV, development of cognitive impairment, and changes in response to herpes viruses (anti-CMV and anti-EBV) over 24 months of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zivadinov, MD, PhD, Principal Investigator — SUNY University at Buffalo
Locations (1):
- Buffalo Neuroimaging Analysis Center, Buffalo, New York, United States